CLINICAL TRIAL: NCT00001248
Title: Evaluation of Progression in Multiple Sclerosis by Magnetic Resonance Imaging (MRI)
Brief Title: Magnetic Resonance Imaging (MRI) to Evaluate Activity of Multiple Sclerosis (MS)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890045; 89-N-0045
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MRI (Magnetic Resonance Imaging); Natural History
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers: Healthy volunteers for technique development and comparison with the patient populations.
- MS/CIS/RIS population: Patients with a diagnosis of MS or who have typical imaging abnormalities associated with MS.
- Non-MS comparison population: Patients with disorders of the CNS, to include patients with diseases that share mechanisms of tissue damage with MS

SUMMARY:
Studies performed under 89-N-0045 are designed to examine the natural history of multiple sclerosis (MS) using MRI and immunological measures. In addition to studying the natural history of untreated patients, the natural history of patients receiving approved disease-modifying therapies of MS will be examined. In both cohorts of patients levels of disease activity on MRI will be compared with immunological characteristics in order to help identify disease mechanism. Patients with either definite MS (based either on clinical or combined clinical and MRI criteria) or with an initial presentation of neurological dysfunction consistent with MS will be studied longitudinally by MRI. Disease activity on MRI will be assessed using several MRI measures of disease activity including the number of contrast enhancing lesions, the overall burden of disease, brain atrophy and measures to assess axonal damage. Patients will be assessed clinically and correlations between immunological and genetic factors and disease activity as seen clinically or by MRI will be studied.

A second cohort of patients starting the use of approved therapy will also be examined. Patients referred to NIH prior to beginning approved therapy will be assessed with a series of three monthly MRIs to determine the level of pretreatment disease activity. After beginning approved therapy under the direction of their private physician, patients will be followed similarly to the natural history cohort. Immunological and genetic findings will be accessed before and during therapy in order to help establish the mechanisms of action of the therapies and to identify mechanisms accounting for either a response or lack of response to therapy. Part of the collected samples willl be cryopreserved to provide respository for further studies focusing on detection of biomarkers indicative of disease state, disease stage or repsonse to therapies.

Additionally, a cohort of normal volunteers will be studied. The studies in the normal volunteers will be used to establish the most appropriate imaging sequences for studying normal white matter in MS patients using magnetization transfer (MT) imaging sequences for studying normal white matter in MS patients using magnetization transfer (MT) imaging and to provide normative immunological measures.

DETAILED DESCRIPTION:
Study Description:

This study is primarily designed to examine the evolving natural history of multiple sclerosis (MS) and its mimickers, viewed through the window of neuroimaging (especially magnetic resonance imaging or MRI). After required baseline evaluation, follow-up study timepoints are driven by clinical standard-of-care, and data from clinically driven procedures may be analyzed for research. Optional research procedures may also be performed during these visits. Optional research-only visits may be scheduled to further investigate findings from the clinical visits. The same research procedures may be performed in healthy volunteers to assess whether the research findings are specific to the affected participant group.

Objectives:

To describe the evolving natural history of MS, viewed clinically, radiologically, and biologically, both prior to and after the introduction of increasingly effective disease modifying therapies (DMT). The protocol has three other important objectives: (1) screening prospective participants for selected NINDS Neuroimmunology Clinic trials; (2) studying healthy volunteers for comparison with affected participants and for development of new experimental technologies; and (3) comparing MS to other neurological diseases that share imaging or clinical features.

Endpoints:

The primary endpoint is the rate of change in the number of new white matter lesions per participant, indexed by the date of baseline evaluation.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. One of the following:

   1. Affected participant with either a diagnosis of MS based on currently accepted diagnostic criteria, or imaging or clinical abnormalities associated with MS.
   2. Healthy volunteer.
2. Age >=18
3. Able to give informed consent.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Contraindication to MRI at the time of initial enrollment (with the exception of pregnancy).
2. Unwilling to allow coded samples to be processed offsite or unwilling to have coded samples used in other studies.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: -MS/CIS/RIS population-Patients with a diagnosis of MS or who have typical imaging abnormalities associated with MS.-Non-MS comparison populations-Patients with disorders of the CNS, to include patients with diseases that share mechanisms of tissue damage with MS, such as mitochondrial disorders, leukodystrophies, neurodegenerative diseases that may cause axonal loss or oxidative stress, and chronic small vessel disease.-Healthy volunteers-Healthy volunteers for technique development and comparison with the patient populations.
Sampling Method: Non-Probability Sample
Enrollment: 3750 (Estimated)
Dates: Start 1992-07-23 (Actual)

PRIMARY OUTCOMES:
the rate of change in the number of new white matter lesions per participant | baseline vs. follow up visits
  The primary outcome, which is designed to determine how MS disease activity has changed with the advent of ever-more-effective disease-modifying therapy, is the rate of change in the number of new white matter lesions per participant, indexed by the date of baseline evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a natural history, not a clinical trial, therefore we are not obligated to provide a data sharing statement.

REFERENCES:
- [Background] Tresley RM, Stone LA, Fields N, Maloni H, McFarland H, Frank JA. Clinical safety of serial monthly administrations of gadopentetate dimeglumine in patients with multiple sclerosis: implications for natural history and early-phase treatment trials. Neurology. 1997 Apr;48(4):832-5. doi: 10.1212/wnl.48.4.832. PMID 9109864
- [Background] Calabresi PA, Stone LA, Bash CN, Frank JA, McFarland HF. Interferon beta results in immediate reduction of contrast-enhanced MRI lesions in multiple sclerosis patients followed by weekly MRI. Neurology. 1997 May;48(5):1446-8. doi: 10.1212/wnl.48.5.1446. PMID 9153489
- [Background] Calabresi PA, Tranquill LR, Dambrosia JM, Stone LA, Maloni H, Bash CN, Frank JA, McFarland HF. Increases in soluble VCAM-1 correlate with a decrease in MRI lesions in multiple sclerosis treated with interferon beta-1b. Ann Neurol. 1997 May;41(5):669-74. doi: 10.1002/ana.410410517. PMID 9153530
- [Derived] Al-Louzi O, Letchuman V, Manukyan S, Beck ES, Roy S, Ohayon J, Pham DL, Cortese I, Sati P, Reich DS. Central Vein Sign Profile of Newly Developing Lesions in Multiple Sclerosis: A 3-Year Longitudinal Study. Neurol Neuroimmunol Neuroinflamm. 2022 Jan 13;9(2):e1120. doi: 10.1212/NXI.0000000000001120. Print 2022 Mar. PMID 35027474
- [Derived] Absinta M, Sati P, Schindler M, Leibovitch EC, Ohayon J, Wu T, Meani A, Filippi M, Jacobson S, Cortese IC, Reich DS. Persistent 7-tesla phase rim predicts poor outcome in new multiple sclerosis patient lesions. J Clin Invest. 2016 Jul 1;126(7):2597-609. doi: 10.1172/JCI86198. Epub 2016 Jun 6. PMID 27270171
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1989-N-0045.html